CLINICAL TRIAL: NCT00729469
Title: Efficacy and Safety of Ospemifene in the Treatment of Moderate to Severe Vaginal Dryness and Vaginal Pain Associated With Sexual Activity, Symptoms of Vulvar and Vaginal Atrophy (VVA), Associated With Menopause: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing Oral Ospemifene 60 mg Dose With Placebo in Postmenopausal Women
Brief Title: Efficacy and Safety of Ospemifene in the Treatment of Moderate to Severe Vaginal Dryness and Vaginal Pain Associated With Sexual Activity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Collaborators: Hormos Medical (Industry); QuatRx Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-50821
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Atrophy; Vaginal Diseases
Keywords: Vulvar and vaginal atrophy in postmenopausal women; Menopausal symptoms; Vaginal atrophy; Urogenital atrophy
MeSH Terms: conditions — Atrophy; Vaginal Diseases | interventions — Ospemifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Ospemifene 60 mg/day and K-Y® lubricant (Experimental): Subjects will receive a single, oral dose (1 tablet) of ospemifene 60 mg each morning with food for 12 weeks. All subjects will be provided vaginal lubricant (K-Y® Brand) and should use it as needed.
  Interventions: Drug: Ospemifene 60 mg
- Placebo and K-Y® lubricant (Placebo Comparator): Subjects will receive a single, oral dose (1 tablet) of Placebo each morning with food for 12 weeks. All subjects will be provided vaginal lubricant (K-Y® Brand) and should use it as needed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ospemifene 60 mg — 60 mg/day oral dose of ospemifene for 12 weeks - from Visit 2 (Randomization, Day 1) to Visit 4 (Week 12) plus Non-hormonal vaginal lubricant as needed
  Other Names: Osphena®
  Arms: Ospemifene 60 mg/day and K-Y® lubricant
Drug: Placebo — oral dose of placebo,1 tablet/day, for 12 weeks - from Visit 2 (Randomization, Day 1) to Visit 4 (Week 12) plus Non-hormonal vaginal lubricant as needed
  Arms: Placebo and K-Y® lubricant

SUMMARY:
The purpose of this study is to determine the safety and efficacy of ospemifene in postmenopausal women experiencing moderate to severe vaginal dryness and vaginal pain associated with sexual activity.

ELIGIBILITY:
Inclusion Criteria:

* Naturally or surgically menopausal
* Moderate or severe symptoms of vaginal atrophy
* 5% or fewer superficial cells in maturation index of vaginal smear
* Vaginal pH greater than 5.0
* Self reported Most Bothersome Symptom of vaginal dryness or vaginal pain associated with sexual activity, with a severity of moderate or severe at randomization

Exclusion Criteria:

* Uterine bleeding of unknown origin, uterine polyps or symptomatic and/or large uterine fibroids
* Current vaginal infection requiring medication
* Clinically significant abnormal gynecological findings other than signs of vaginal atrophy (e.g.

uterine or vaginal prolapse of Grade 2 or higher)

* Previous participation in any other ospemifene study

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 919 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

REFERENCES:
- [Derived] Portman DJ, Bachmann GA, Simon JA; Ospemifene Study Group. Ospemifene, a novel selective estrogen receptor modulator for treating dyspareunia associated with postmenopausal vulvar and vaginal atrophy. Menopause. 2013 Jun;20(6):623-30. doi: 10.1097/gme.0b013e318279ba64. PMID 23361170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was screened on August 04, 2008 and last patient completed on July 30, 2009
Pre-assignment Details: Subjects reporting moderate to severe VVA symptoms of vaginal dryness or vaginal pain associated with sexual activity as the most bothersome symptom (MBS) at the initial screening visit were allowed to continue in the screening phase of the study. Each subject entered 1 of 2 strata based on their self-reported moderate to severe MBS
Groups:
- Subjects on Placebo: Subjects received a single, oral dose (1 tablet) of placebo each morning with food for 12 weeks. All subjects were provided with vaginal lubricant (K-Y® Brand), which was used as needed.
- Subjects on Ospemifene 60 mg/Day: Subjects received a single, oral dose (1 tablet) of ospemifene 60 mg each morning with food for 12 weeks. All subjects were provided with vaginal lubricant (K-Y® Brand), which was used as needed.
Period: Overall Study
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Started | 456 | 463
Completed | 403 | 416
Not Completed | 53 | 47
Not completed — Adverse Event | 14 | 25
Not completed — Lost to Follow-up | 9 | 9
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 19 | 8
Not completed — Other-Not mentioned | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day | Total
Number analyzed (Participants) | 456 | 463 | 919
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (6.39) | 58.7 (6.56) | 58.6 (6.47)
Age, Customized [Number; unit: participants]
  <45 | 7 | 8 | 15
  45-54 | 106 | 113 | 219
  55-64 | 266 | 260 | 526
  >=65 | 77 | 82 | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 456 | 463 | 919
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 396 | 409 | 805
  Black or African American | 35 | 28 | 63
  Asian | 3 | 8 | 11
  Pacific Islander | 0 | 2 | 2
  Other | 22 | 16 | 38
Height [Mean (Standard Deviation); unit: cm] | 162.6 (6.39) | 162.3 (6.34) | 162.5 (6.36)
Weight [Mean (Standard Deviation); unit: kg] | 69.38 (12.38) | 68.98 (12.38) | 69.18 (12.37)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.21 (4.32) | 26.16 (4.31) | 26.18 (4.31)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Percentage of Parabasal Cells in the Maturation Index of the Vaginal Smear (Dryness Strata)
Time Frame: 12 weeks
Population: ITT; LOCF
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 154 | 160
percentage of parabasal cells | -3.7 (29.97) | -31.7 (37.25)

2. Primary Outcome: Change From Baseline to Week 12 in Percentage of Superficial Cells in the Maturation Index of the Vaginal Smears (Dryness Strata)
Time Frame: 12 weeks
Population: ITT; LOCF
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 154 | 160
percentage of superficial cells | 3.3 (9.02) [-11 to 57] | 12.4 (15.36) [-4 to 65]

3. Primary Outcome: Change From Baseline to Week 12 in Vaginal pH (Dryness Strata)
Time Frame: 12 weeks
Population: ITT; LOCF
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 154 | 160
pH | -0.24 (0.800) | -0.92 (1.100)

4. Secondary Outcome: Change From Baseline to Week 4 in Percentage of Parabasal Cells in the Maturation Index (Dryness Strata)
Time Frame: 4 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 154 | 160
percentage of parabasal cells | -2.8 (2.18) | -31.2 (2.15)

5. Secondary Outcome: Change From Baseline to Week 4 in Percentage of Superficial Cells in the Maturation Index (Dryness Strata)
Time Frame: 4 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 154 | 160
percentage of superficial cells | 3.6 (1.07) | 12.7 (1.05)

6. Primary Outcome: Change From Baseline to Week 12 in Severity of the Most Bothersome Symptom of Vaginal Dryness Associated With Sexual Activity (Dryness Strata)
Time Frame: 12 weeks
Population: ITT; LOCF
Measure: Number; unit: participants
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 154 | 160
participants
  -3 (Sev. to none) | 14 | 23
  -2 (Sev. to mild, or mod. to none) | 39 | 51
  -1 (Sev. to mod., mod.to mild, or mild to none) | 52 | 39
  0 (No change) | 44 | 44
  1 (None to mild, mild to mod., or mod. to sev.) | 5 | 3

7. Primary Outcome: Change From Baseline to Week 12 in Percentage of Parabasal Cells in the Maturation Index of the Vaginal Smear (Dyspareunia Strata)
Time Frame: 12 weeks
Population: ITT; LOCF
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 302 | 303
percentage of parabasal cells | 0.0 (30.00) | -40.2 (38.80)

8. Primary Outcome: Change From Baseline to Week 12 in Percentage of Superficial Cells in the Maturation Index of the Vaginal Smears (Dyspareunia Strata)
Time Frame: 12 weeks
Population: ITT; LOCF
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 302 | 303
percentage of superficial cells | 1.7 (6.88) | 12.3 (14.77)

9. Primary Outcome: Change From Baseline to Week 12 in Vaginal pH (Dyspareunia Strata)
Time Frame: 12 weeks
Population: ITT; LOCF
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 302 | 303
pH | -0.07 (0.814) | -0.94 (1.016)

10. Primary Outcome: Change From Baseline to Week 12 in Severity of the Most Bothersome Symptom of Vaginal Pain Associated With Sexual Activity (Dyspareunia Strata)
Time Frame: 12 weeks
Population: ITT; LOCF
Measure: Number; unit: participants
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 302 | 303
participants
  -3 (Sev. to none) | 47 | 67
  -2 (Sev. to mild, or mod. to none) | 70 | 93
  -1 (Sev. to mod., mod.to mild, or mild to none) | 76 | 82
  0 (No change) | 102 | 55
  1 (None to mild, mild to mod., or mod. to sev.) | 7 | 6

11. Secondary Outcome: Change From Baseline to Week 4 in Vaginal pH (Dryness Strata)
Time Frame: 4 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 154 | 160
pH | -0.21 (0.884) | -0.81 (0.962)

12. Secondary Outcome: Change From Baseline to Week 4 in Severity of Most Bothersome Symptom of Vaginal Dryness Associated With Sexual Activity (Dryness Strata)
Time Frame: 4 weeks
Population: ITT; change from baseline to week 4 in severity of most bothersome symptom of vaginal dryness associated with sexual activity (dryness strata) was assessed in 152 subjects in the placebo group and 154 subjects in the ospemifene 60 mg/day group.
Measure: Number; unit: participants
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 152 | 154
participants
  -3 (Sev. to None) | 9 | 11
  -2 (Sev. to Mild, or Mod. to None) | 25 | 31
  -1 (Sev. to Mod., Mod. to Mild, or Mild to None) | 57 | 67
  0 (No change) | 60 | 40
  1 (None to Mild, Mild to Mod., or Mod. to Sev.) | 1 | 5

13. Secondary Outcome: Change From Baseline to Week 4 in Vaginal pH (Dyspareunia Strata)
Time Frame: 4 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 302 | 303
pH | -0.15 (0.821) | -0.82 (0.979)

14. Secondary Outcome: Change From Baseline to Week 4 in Severity of Most Bothersome Symptom of Vaginal Pain Associated With Sexual Activity (Dyspareunia Strata)
Time Frame: 4 weeks
Population: ITT; change from baseline to week 4 in severity of most bothersome symptom of vaginal pain associated with sexual activity (dyspareunia strata) was assessed in 287 subjects in the placebo group and 295 subjects in the ospemifene 60 mg/day group.
Measure: Number; unit: participants
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 287 | 295
participants
  -3 (Sev. to None) | 34 | 39
  -2 (Sev. to Mild, or Mod. to None) | 64 | 72
  -1 (Sev. to Mod., Mod. to Mild, or Mild to None) | 84 | 97
  0 (No change) | 95 | 78
  1 (None to Mild, Mild to Mod., or Mod. to Sev.) | 10 | 9

15. Secondary Outcome: Change From Baseline to Week 4 in Percentage of Parabasal Cells in the Maturation Index (Dyspareunia Strata)
Time Frame: 4 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 302 | 303
percentage of parabasal cells | -0.8 (1.59) | -37.8 (1.54)

16. Secondary Outcome: Change From Baseline to Week 4 in Percentage of Superficial Cells in the Maturation Index (Dyspareunia Strata)
Time Frame: 4 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Number analyzed (Participants) | 302 | 303
percentage of superficial cells | 1.9 (0.69) | 13.0 (0.67)

ADVERSE EVENTS:
Time Frame: 16 Weeks During the time period after the signing of the informed consent form and including the collection of the last safety information
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 60 mg/Day
Serious Adverse Events (participants affected / at risk) | 7/456 | 6/463
Other Adverse Events (participants affected / at risk) | 102/456 | 153/463
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects on Placebo (N=456) | Subjects on Ospemifene 60 mg/Day (N=463)
Palpitations (Cardiac disorders) | 1 | 0
Autoimmune Thyroiditis (Endocrine disorders) | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2
Peridiverticular Abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial Aneurysm (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Bipolar Disorder (Psychiatric disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0
Bladder Prolapse (Renal and urinary disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects on Placebo (N=456) | Subjects on Ospemifene 60 mg/Day (N=463)
Urinary Tract Infection (Infections and infestations) | 23 | 37
Nasopharyngitis (Infections and infestations) | 16 | 20
Vulvovaginal Candidiasis (Infections and infestations) | 2 | 18
Vulvovaginal Mycotic Infection (Infections and infestations) | 2 | 17
Upper Respiratory Tract Infection (Infections and infestations) | 21 | 15
Sinusitis (Infections and infestations) | 25 | 11
Headache (Nervous system disorders) | 21 | 16
Vaginal Discharge (Reproductive system and breast disorders) | 3 | 21
Hot Flush (Vascular disorders) | 15 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.